CLINICAL TRIAL: NCT03070691
Title: A Randomized, Double-blind, Vehicle-controlled, Multicenter Trial of Topically Administered LDE225 Cream (0.75% Bid) to Evaluate Clearance of Basal Cell Carcinoma in Adult Patients With Nevoid Basal Cell Carcinoma Syndrome
Brief Title: Efficacy, Safety and Tolerability of Topically Applied LDE225 Cream (Hedgehog Pathway Inhibitor) in Adult Patients With Nevoid Basal Cell Carcinoma Syndrome (NBCCS)
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLDE225B2307
Record Dates: First submitted 2010-07-06; First posted 2017-03-03 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-02

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal cell carcinoma; Nevoid Basal Cell Carcinoma Syndrome; NBCCS, Gorlin syndrome; Gorlin-Goltz Syndrome; Basal Cell Nevus Syndrome; BCNS, Hedgehog pathway inhibitor; topical; Smoothened
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDE225 0.75% cream (Active Comparator)
  Interventions: Drug: LDE225B
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: LDE225B — Cream, 2x daily
  Arms: LDE225 0.75% cream
Drug: Vehicle — cream, 2x daily
  Arms: Vehicle

SUMMARY:
This 22 week study will assess the efficacy, safety, and tolerability of LDE225 versus vehicle when applied topically to basal cell carcinoma (BCC) in patients with NBCCS. Patients will treat multiple BCCs for up to 12 weeks. Treatment success is defined as complete clinical clearance and complete histological clearance in BCCs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult greater than 18 years old, male or female.
2. Patient must be able to understand and communicate with the investigator and comply with the requirements of the study.
3. Typical presentation of NBCCS in the opinion of the investigator
4. At least one of the major clinical criteria of NBCCS.
5. Multiple BCCs during the screening period

Exclusion Criteria:

1. Any concomitant dermatological disease that could confound the evaluations, based on the discretion of the investigator.
2. Prior exposure to LDE225.
3. Use of systemic treatment for BCC in the 4 weeks prior to Baseline.
4. Use of topical treatment or photodynamic therapy (PDT) in the 12 weeks prior to Baseline.
5. Use of other investigational drugs at Baseline, or within 30 days or 5 half-lives prior to Baseline, whichever is longer.
6. Clinically significant medical condition, as per judgment of the investigator.
7. History of hypersensitivity to any of the ingredient of the study drug.
8. Pregnant or nursing (lactating) women
9. Women of child-bearing potential and fertile males, UNLESS they are using two birth control methods

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To demonstrate superiority of topical LDE225 versus vehicle in terms of treatment success in patients with NBCCs. Measure: Complete clinical clearance and complete histological clearance of BCCs | 4 weeks after LDE225 treatment

SECONDARY OUTCOMES:
To assess the safety of topical treatment with LDE225, compared to vehicle. Measure: Reported systemic adverse events in patients with NBCCS | Treatment phase and up to 4 weeks after LDE225 treatment
To evaluate the local tolerability of topical treatment with LDE225, compared to vehicle. Measure:Reported local adverse events in patients with NBCCS | Treatment phase and up to 4 weeks after LDE225 treatment
To assess the rate of complete clinical clearance of BCCs in patients with NBCCS. Measure: No clinical residual signs of carcinoma | 4 weeks after LDE225 treatment
To assess the rate of complete histological clearance of BCCs in patients with NBCCS. Measure: No residual tumor tissue | 4 weeks after LDE225 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- Belgium (2):
  - Novartis Investigative site, Brussels
  - Novartis Investigative site, Leuven
- Canada (2):
  - Novartis Investigative site, Waterloo, Ontario
  - Novartis Investigative site, Sainte-Foy, Quebec
- Novartis Investigative site, Prague, Czechia
- Novartis Investigative site, Helsinki, Finland
- Germany (15):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Munich
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Würzburg
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative site, Thessaloniki
- Italy (5):
  - Novartis Investigative site, Catania
  - Novartis Investigative site, L’Aquila
  - Novartis Investigative site, Napoli
  - Novartis Investigative site, Padua
  - Novartis Investigative site, Siena
- Spain (2):
  - Novartis Investigative site, Barcelona
  - Novartis Investigative site, Madrid
- Switzerland (2):
  - Novartis Investigative site, Lausanne
  - Novartis Investigative site, Zurich
- United Kingdom (3):
  - Novartis Investigative site, Glasgow
  - Novartis Investigative site, London
  - Novartis Investigative site, Manchester